CLINICAL TRIAL: NCT03665480
Title: The Effect of Granulocyte-colony Stimulating Factor (G-CSF) on Minimal Residual Disease (MRD) After Induction Therapy in Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: The Effect of G-CSF on MRD After Induction Therapy in Newly Diagnosed AML
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G-CSF on MRD in AML
Record Dates: First submitted 2018-08-07; First posted 2018-09-11 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Granulocyte Colony-stimulating Factor; Minimal Residual Disease; Acute Myeloid Leukemia
MeSH Terms: conditions — Neoplasm, Residual; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF treatment (Experimental): In G-CSF treatment group, all participants are treated with G-CSF at the dose of 5ug/kg per day until neutrophil higher than 0.5 g/L or 14 days from day three after induction therapy. MRD is monitored at day 14 and 28 with flow cytometry and quantity PCR if a fusion gene is available.
  Interventions: Drug: G-SCF
- G-CSF-free (No Intervention): In G-CSF-free group, no participants with newly diagnosed AML are treated with G-CSF after induction therapy.

INTERVENTIONS:
Drug: G-SCF — In G-CSF treatment group, all patients are treated with G-CSF at the dose of 5ug/kg pre day until neutrophil higher than 0.5 g/L or 14 days from day three after induction therapy. MRD is monitored at day 14 and 28, respectively, with flow cytometry and quantity PCR if a fusion gene is available.
  Arms: G-CSF treatment

SUMMARY:
Granulocyte-colony stimulating factor (G-CSF) is konwn to have no significant effect on leukemia stem cells and has been widely used in the patients with agranulocytosis after chemotherapy. Minimal residual disease (MRD), an index for early treatment response, plays an important role in prognostic prediction. Numbers of data have shown MRD at day 14 after induction therapy significantly predicts prognosis. However, the retrospetive data from the investigators showed that patients with G-CSF treatment after induction had higher MRD at day 14 but not significantly different at day 28, suggesting that G-CSF might work on the differenciation of hemapoetic stem cells and increase MRD levels at day 14. In this multicenter prospective randomized controlled study, the effect of G-CSF on MRD after induction therapy in newly diagnosed acute myeloid leukemia (AML) is evaluated.

DETAILED DESCRIPTION:
Granulocyte-colony stimulating factor (G-CSF) is konwn to have no significant effect on leukemia stem cells and has been widely used in the patients with agranulocytosis after chemotherapy. Minimal residual disease (MRD), an good index for early treatment response, plays an important role in prognostic prediction. Numbers of data have shown MRD at day 14 after induction therapy significantly predicts prognosis. However, the retrospetive data from the investigators showed that patients with G-CSF treatment after induction had higher MRD at day 14 but not significantly different at day 28,suggesting that G-CSF might work on the differenciation of hemapoetic stem cells and increase MRD level at day 14. In this multicenter prospective study, the investigators randomizedly divide all participants with newly diagnosed acute myeloid leukemia (AML) into G-CSF treatment group and G-SCF-free group. In G-CSF treatment group, all participants are treated with G-CSF at the dose of 5ug/kg pre day until neutrophil higher than 0.5 g/L or 14 days from day three after induction therapy. MRD is monitored at day 14 and 28 with flow cytometry and quantity PCR if a fusion gene is available in both G-CSF treatment and G-CSF-free groups. Comparision of the difference of MRD levels between the two groups is performed to evaluate the effect of G-CSF on MRD.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed AML exclusively of APL; 14-65 years old; Neutrophil < 1.5 G/L at the day three after induction.

Exclusion Criteria:

Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure); Patients with any conditions not suitable for the trial; NR at day 28 after induction.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
MRD1 | Day 14 after induction
  MRD level is detested by flow cytometry at the day 14 after induction therapy.

SECONDARY OUTCOMES:
OS rate | 2 years
  OS is the abbreviation of overall survival. OS rate is caculated as the ratio of survival participants versus total participants during the 2-year follow-up after diagosis.
DFS rate | 2 years
  DFS is the abbreviation of disease-free survival. DFS rate is caculated as the ratio of participants with continuous complete remission (CR) versus total participants abtaining CR after induction during the 2-year follow-up after diagosis.
Time for neutropenia | 30 days after induction
  The lasting time for the patients with neutropenia after induction therapy
Infection incidence | 30 days after induction
  The incidence of infection after induction
MRD2 | Day 28 after induction
  MRD level is detested by flow cytometry at the day 28 after induction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China